CLINICAL TRIAL: NCT01162616
Title: Is There a Dose-dependant Effect of Sorghum Polyphenols on Human Iron Absorption and Can it be Overcome by Sodium Iron EDTA or by Adding Vitamin C or Laccase?
Brief Title: Polyphenols in Sorghum and Iron Absorption
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Msc, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PP_Fe_Study Sorghum
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Iron Absorption in Presence of Polyphenols
Keywords: iron absorption; polyphenols; sodium iron EDTA; sorghum

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Iron absorption (Other)
  Interventions: Dietary Supplement: labeled iron solutions

INTERVENTIONS:
Dietary Supplement: labeled iron solutions — labeled iron as 2 mg 58FeSO4, 57FeSO4 or 54FeSO4 per test portion (50g sorghum) 2 mg labeled iron as NaFeEDTA per test portion (50g sorghum)

SUMMARY:
Iron deficiency and iron deficiency anemia are two major public health problems in developing countries. In these countries, the use of monotonous plant-based diets, low in animal source food but high in iron absorption inhibitors such as phytic acid or polyphenol, lead to poor iron status or aggravate poor iron status caused by infections. In many West African countries sorghum is a major source of energy, protein, vitamins and minerals especially for the most poverty-stricken people. Some sorghum varieties are known to contain high levels of polyphenols which have an inhibitory effect on iron absorption in humans. Polyphenols are a huge group of plant metabolites with varying chemical structures. Depending on their structure, the level of complex formation with iron in the intestine and thus the negative effect on iron absorption is different.

Micronutrient deficiency can be combated by fortification of plant-based staples. Fortification is a promising food-based approach which can be applied when other strategies fail to provide adequate levels of the respective micronutrient in the diet. To fortify foods with iron, a wide variety of different iron compounds have been used. The iron compound sodium iron ethylenediaminetetraacetic (NaFeEDTA) overcomes the inhibitory effect of phytate on human iron absorption. No information about the potential enhancing effect of NaFeEDTA in presence of polyphenol is available.

The aims of the study are to investigate the effect of different sorghum polyphenol concentrations on human iron absorption and to investigate if the negative impact of the polyphenols can be overcome by using NaFeEDTA as iron compound. The study will include 32 apparently healthy young women which will consume sorghum porridges with different polyphenol levels and sorghum porridges fortified with ferrous sulfate as compared to NaFeEDTA. Furthermore test meals with added vitamin C or added laccase will be compared to a control meal. Iron absorption will be determined by stable isotope technique.

ELIGIBILITY:
Inclusion Criteria:

* Females of reproductive age, 18-40 years
* Maximum body weight 65 kg
* Normal body mass index (18.5-25 kg/m2)
* No intake of mineral/vitamin supplements 2 weeks before and during the study
* No metabolic or gastrointestinal disorders

Exclusion Criteria:

* Pregnancy or lactation
* Regular intake of medication (except oral contraceptives)
* Blood donation or significant blood loss (accident, surgery) over the past 4 months
* Currently participating in another clinical trial or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Former participation in a study involving administration of iron stable isotopes
* Subject who cannot be expected to comply with study protocol
* Eating disorders or food allergy
* High C-reactive protein levels (>5 mg/L)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Iron isotope ratio in blood samples | Study day 17 (16 days after administration of isotopic label in the first test meal/End of the study)
  Whole blood samples will be collected to measure the shift in iron isotope ratios 16 days after administration of isotopic label in the first test meal.
  First test meal on study day 1, Second test meal on study day 2, Third (last) test meal on study day 3, Measurement of iron isotopic shift in blood samples collected on study day 17

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, Prof., Principal Investigator — Swiss Federal Institute of Technology (ETH Zürich)
Locations (1):
- Swiss Federal Institute of Technology ETH Zurich, Zurich, Canton of Zurich, Switzerland